CLINICAL TRIAL: NCT06375577
Title: Evaluating the Speed of Carbohydrate Supplement Absorption in an Athletic Population
Brief Title: Speed of Glucose Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Dr. Chris Gaffney, Senior Lecturer in Integrative Physiology, Lancaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LMS-24-Dean-1
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-08

CONDITIONS: Healthy; Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: This will be a double-blind randomised crossover design. There will be 1 group of participants who will complete all three conditions at random:
  Condition 1 - consume Voom Pocket Rocket. Condition 2 - consume SIS Isotonic Energy Gel. Condition 3 - consume Maurten Gel 160.
  All participants will undergo the same measures - blood sampling for blood glucose, blood lactate, electrolytes and insulin, and monitoring of gas exchange during each study visit.
Who Masked: Participant, Investigator
Masking Description: Both the participants and investigators will be blinded to what supplement they are consuming on each visit. Each supplement will taste the same, and be placed into identical packaging, and be randomly labelled (e.g., A, B, C). This will be done to avoid potential bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Voom Pocket Rocket Electro Energy Bar (Experimental): After at least a 1 week washout period, every participant will undergo a different intervention
  Interventions: Dietary Supplement: 45 grams Voom Pocket Rocket Electro Energy
- Maurten gel 160 (Experimental): After at least a1 week washout period, every participant will undergo a different intervention
  Interventions: Dietary Supplement: 45 grams Maurten Gel 160
- SIS Go isotonic Gel (Experimental): After at least 1 week washout period, every participant will undergo a different intervention
  Interventions: Dietary Supplement: 45 grams SIS Go Isotonic Energy Gel

INTERVENTIONS:
Dietary Supplement: 45 grams Voom Pocket Rocket Electro Energy — Participants will be required to consume 45 grams (in carbohydrates) of the Voom Pocket Rocket Electro Energy on one of the three experimental visits. Participants will have blood glucose, blood lactate, and insulin sampled throughout a 1-hour modified oral glucose tolerance test. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: Voom Pocket Rocket Electro Energy Bar
Dietary Supplement: 45 grams SIS Go Isotonic Energy Gel — Participants will be required to consume 45 grams (in carbohydrates) SIS Isotonic Energy Gel on one of the three experimental visits. Participants will have blood glucose, blood lactate, and insulin sampled throughout a 1-hour modified oral glucose tolerance test. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: SIS Go isotonic Gel
Dietary Supplement: 45 grams Maurten Gel 160 — Participants will be required to consume 45 grams (in carbohydrates) Maurten Gel 160 on one of the three experimental visits. Participants will have blood glucose, blood lactate, and insulin sampled throughout a 1-hour modified oral glucose tolerance test. Gas exchange will also be monitored throughout the 1-hour study visit.
  Arms: Maurten gel 160

SUMMARY:
The purpose of this study is to look at how fast commercially available supplements containing carbohydrate can get into the bloodstream. If carbohydrate, in the form of glucose, gets into the blood faster, this can provide an instant energy source and help fuel the body during exercise. We will be testing three supplements, namely Voom Pocket Rocket, SIS Go Isotonic Energy Gel, and Maurten Gel 160. Each participant will complete all three conditions, consuming one of each supplement at random per condition. The study requires participation from male runners, cyclists and triathletes who are aged between 18-35.

Each visit will take approximately 1 hour and 30 minutes, and three experimental visits per participant. The study will involve frequent blood sampling and the continuous monitoring of gas exchange (oxygen/carbon dioxide). Blood sampling via cannulation will be used to analyse the lactate, glucose, and insulin content of the blood. Gas exchange will measure the oxygen breathed in and carbon dioxide breathed out throughout the study.

The investigators plan to carry out the study on 16 participants who will be a mix of male runners, cyclists and triathletes.

DETAILED DESCRIPTION:
The aim of this study is to investigate and compare the speed of delivery of three commercially available carbohydrate supplements during a 1 hour modified glucose tolerance test. This study will be a randomised double-blind crossover in design. Participants will be required to attend the Human Performance Laboratory at Lancaster University on three separate visits. During each visit, participants will be required to consume one of three commercially available carbohydrate supplements, namely Maurten Gel 160 (MAU), Voom Pocket Rocket Electro Energy Bar (PR), and SIS Go Isotonic Energy Gel (SIS). Each consumable will be blinded to both the researchers and participants, flavoured the same (lemon and lime) and placed into identical packaging with anonymised labelling to minimise the risk of bias. The supplements will be matched for carbohydrate content (45 grams). Blinding of supplements will be completed offsite by people not in the research team and followed strict food and hygiene protocols. Each participant will complete all three conditions, consuming one of each supplement at random per condition.

Each visit will involve frequent venous blood sampling for glucose, lactate and insulin. An anterograde venous cannula will be inserted into a vein in the antecubital fossa of the arm by a qualified member of the research team. This is a less invasive alternative to an arterial cannula whilst still allowing for accurate metabolic measures to be taken. This method is also less painful than inserting a retrograde cannula which can cause significant discomfort.

Once the anterograde venous cannula is inserted and secured in place, a resting measurement of blood will be taken (1ml of blood taken to measure glucose and lactate, and 3ml for insulin). Participants will then be required to consume one of the three carbohydrate energy supplements. Once the supplement had been consumed, continuous gas analysis will begin to analyse gas exchange to non-invasively measure substrate utilisation. This signals the start of the test, and a timer will be set for 1 hour.

Throughout the test, blood sampling will be taken in frequent intervals. 1ml of blood sampled every 5 minutes to check for glucose and lactate, and 3ml of blood sampled every 10 minutes for insulin. Gas exchange will be continuously measured to non-invasively measure substrate utilization in the muscle via indirect calorimetry which determines energy expenditure by measuring the body's oxygen consumption and carbon dioxide production. The measurement is based on the assumption that the volume of oxygen (VO2) consumed is used to oxidise fuels, and the volume of carbon dioxide (VCO2) produced is a by-product of substrate utilisation.

After the study visit, analysis will be conducted assessing how each of the three supplements effect blood glucose, blood lactate, insulin, and gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* Males
* Tier 2 runners, cyclists, and triathletes; local level representation, training ~ 3 times per week, training with a purpose to compete, identify with a specific sport, limited skill development
* BMI between 18.5-24.9 - based on healthy weight range for BMI as per NHS and BMI of recreational to elite long-distance runners

Exclusion Criteria:

* Allergies to any listed ingredients on any supplements.
* Diabetes (type 1 or 2)
* Any medical conditions
* Smokers
* Anyone using drugs or medication
* Anyone consuming alcohol within 24 hours of the study
* Exercise must be restricted within 24 hours of the study
* Caffeine must not be consumed within 24 hours of testing as it can significantly enhance carbohydrate oxidation rates
* Diets including high-carbohydrate-low-fat (HCLF), low-carbohydrate-high-fat (LCHF), ketogenic, and/or glycogen manipulation diets

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only biological males are eligible to participate in this study.
  It was decided that a male only cohort would be included in this study due to the timeframe of the research (undertaken as part of a Masters by Research degree), and that including females would require a larger sample size, and thus a longer timeframe. Research has also found sex differences between responses to glucose absorption, demonstrating that females have a slower glucose absorption time, and that the menstrual cycle can significantly effect glucose absorption which would lengthen the time of research as a greater sample size would be needed with strict controls on contraception & tracking of menstrual cycle.
Enrollment: 16 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Blood Glucose | 1 hour
  Frequent blood sampling for blood glucose (1ml every 5 mins for 1 hour) followed by analysis in the Biosen Analyser
Blood Lactate | 1 hour
  Frequent blood sampling for blood lactate (1ml every 5 mins for 1 hour) followed by analysis in the Biosen Analyser
Insulin | 1 hour
  Frequent blood sampling for insulin (3ml every 10 mins for 1 hour) followed by analysis in an ELISA
Gas Exchange | 1 hour
  Gas exchange measured throughout each 1 hour visit via a Cortex Metalyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Lancaster University, Lancaster, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rauch CE, McCubbin AJ, Gaskell SK, Costa RJS. Feeding Tolerance, Glucose Availability, and Whole-Body Total Carbohydrate and Fat Oxidation in Male Endurance and Ultra-Endurance Runners in Response to Prolonged Exercise, Consuming a Habitual Mixed Macronutrient Diet and Carbohydrate Feeding During Exercise. Front Physiol. 2022 Jan 4;12:773054. doi: 10.3389/fphys.2021.773054. eCollection 2021. PMID 35058795
- [Background] Yeo SE, Jentjens RL, Wallis GA, Jeukendrup AE. Caffeine increases exogenous carbohydrate oxidation during exercise. J Appl Physiol (1985). 2005 Sep;99(3):844-50. doi: 10.1152/japplphysiol.00170.2005. Epub 2005 Apr 14. PMID 15831802
- [Background] Wirnitzer K, Boldt P, Wirnitzer G, Leitzmann C, Tanous D, Motevalli M, Rosemann T, Knechtle B. Health status of recreational runners over 10-km up to ultra-marathon distance based on data of the NURMI Study Step 2. Sci Rep. 2022 Jun 18;12(1):10295. doi: 10.1038/s41598-022-13844-4. PMID 35717392
- [Background] Marc A, Sedeaud A, Guillaume M, Rizk M, Schipman J, Antero-Jacquemin J, Haida A, Berthelot G, Toussaint JF. Marathon progress: demography, morphology and environment. J Sports Sci. 2014;32(6):524-32. doi: 10.1080/02640414.2013.835436. Epub 2013 Nov 5. PMID 24191965
- [Background] Williams PT, Satariano WA. Relationships of age and weekly running distance to BMI and circumferences in 41,582 physically active women. Obes Res. 2005 Aug;13(8):1370-80. doi: 10.1038/oby.2005.166. PMID 16129719
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] Horie I, Abiru N, Eto M, Sako A, Akeshima J, Nakao T, Nakashima Y, Niri T, Ito A, Nozaki A, Haraguchi A, Akazawa S, Mori Y, Ando T, Kawakami A. Sex differences in insulin and glucagon responses for glucose homeostasis in young healthy Japanese adults. J Diabetes Investig. 2018 Nov;9(6):1283-1287. doi: 10.1111/jdi.12829. Epub 2018 Mar 30. PMID 29489067
- [Background] Lin G, Siddiqui R, Lin Z, Blodgett JM, Patel SN, Truong KN, Mariakakis A. Blood glucose variance measured by continuous glucose monitors across the menstrual cycle. NPJ Digit Med. 2023 Aug 11;6(1):140. doi: 10.1038/s41746-023-00884-x. PMID 37567949
- [Background] McGuire EA, Helderman JH, Tobin JD, Andres R, Berman M. Effects of arterial versus venous sampling on analysis of glucose kinetics in man. J Appl Physiol. 1976 Oct;41(4):565-73. doi: 10.1152/jappl.1976.41.4.565. PMID 985402
- [Background] Brooks DC, Black PR, Arcangeli MA, Aoki TT, Wilmore DW. The heated dorsal hand vein: an alternative arterial sampling site. JPEN J Parenter Enteral Nutr. 1989 Jan-Feb;13(1):102-5. doi: 10.1177/0148607189013001102. PMID 2926973
- [Background] Copeland KC, Kenney FA, Nair KS. Heated dorsal hand vein sampling for metabolic studies: a reappraisal. Am J Physiol. 1992 Nov;263(5):E1010-4. doi: 10.1152/ajpendo.1992.263.5.E1010. PMID 1443110
- [Background] Wrench, E., 2021. Determining the Dose-Response Relationship Between Exercise and Glycaemic Control and Examining Exercise as a Treatment for Type 2 Diabetes (Master's thesis, Lancaster University (United Kingdom)).
- [Background] Delsoglio M, Achamrah N, Berger MM, Pichard C. Indirect Calorimetry in Clinical Practice. J Clin Med. 2019 Sep 5;8(9):1387. doi: 10.3390/jcm8091387. PMID 31491883
- See also: Voom Pocket Rocket Electro Energy — https://www.voomnutrition.co.uk/products/pocket-rocket-electro-energy-bar
- See also: SIS Go Isotonic Energy Gel — https://www.scienceinsport.com/shop-sis/go-range/go-gels/sis-go-isotonic-energy-gel-pack
- See also: Maurten Gel 160 — https://www.maurten.com/products/gel-160?gad_source=1&gclid=Cj0KCQjwn7mwBhCiARIsAGoxjaL26EyCLaxZsOcGcyle44lSI_HlwDOZKp2P5-bL7rqMDUAaTObREqgaAvncEALw_wcB